CLINICAL TRIAL: NCT06679010
Title: A Therapist-guided Online-delivered Group Counseling Program for Pregnant Women and New Mothers With ADHD: A Feasibility Study of AMOR; ADHD, Mothers Online Resources
Brief Title: A Feasibility Study of AMOR; ADHD, Mothers Online Resources
Acronym: AMOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Sygeforsikringen danmark (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S-20240074; 2021-0139 (Other Grant/Funding Number: Sygeforsikring Danmark)
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy; Mother; Women; Attention Deficit Disorder With Hyperactivity; Postpartum Depression (PPD); Anxiety; Stress; Emotional Dysregulation; Quality of Life
Keywords: AMOR; feasibility; online counselling of pregnant women with ADHD; mixed methods evaluation
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Depression, Postpartum; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The study is a feasibility trial with an uncontrolled, within-group, pre-post design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental)
  Interventions: Other: Online group counseling

INTERVENTIONS:
Other: Online group counseling — The program progresses as one weekly group session over 10 weeks, each with its own topic. The core components of the program include psychoeducation, training self-compassion and acceptance, cognitive restructuring, interpersonal skills training, systems and management of daily life activities, prevention of conflicts, and the mother-baby relation. Participants will meet online as a group together with the instructor, a consultant from the ADHD Association, who will lead and facilitate the sessions. Before each session, there is a podcast episode that covers the topic of each session. The 10 podcasts feature interviews with clinicians, researchers, and women with ADHD, focusing on the themes from the program's sessions.

SUMMARY:
The primary aim of this study is to investigate the feasibility of the program AMOR for pregnant women and new mothers with Attention Deficit Hyperactivity Disorder (ADHD), by examining adherence, credibility, treatment satisfaction, and negative effects. The secondary objective is to obtain preliminary information about the short-term clinical outcomes of the program on self-report scales assessing symptoms of ADHD, stress, anxiety, depression, difficulties in emotion regulation, and quality of life.

The main questions this study aims to answer:

1. To what extent will pregnant women and new mothers with ADHD adhere to, find useful, be satisfied with, and experience negative effects of the program AMOR?
2. To what extent will pregnant women and new mothers with ADHD experience improvements in ADHD symptoms, stress, anxiety, depression, difficulties in emotion regulation, and quality of life?

Participants will:

* listen to the 10 podcasts in the program
* attend the 10 online guided sessions in the program
* fill in questionnaires related to the primary and secondary objectives
* some will be invited to participate in an online semi-structured interview

DETAILED DESCRIPTION:
Methods The content of the program has been developed by the Danish ADHD Association (ADHD-foreningen) in collaboration with researchers from Aarhus University and the University of Southern Denmark. This program is specifically designed for pregnant women and new mothers with ADHD as an online group intervention. The online format ensures that transportation time is not a barrier to participation, allowing women from across the country to take part. This is particularly important for inclusion, as the program must be accessible during pregnancy. The program is developed based on the extensive knowledge that the ADHD Association has gained from over 40 years of working with people with ADHD. The content is tailored to the key concerns and challenges related to ADHD in the perinatal period, the period related to pregnancy and the first year postpartum and is based on the general principles of cognitive behavioral therapy. It is also inspired by existing literature, a survey among the female members of the ADHD Association, and interviews with women with ADHD about their experiences with pregnancy and postpartum.

Procedure The feasibility trial will be carried out as a mixed-method process evaluation, including both interviews and questionnaire data. The program will proceed over 10 weeks. Questionnaires will be distributed from Research Electronic Data Capture (REDCap) via e-boks at baseline and at 1 week post-program. Interviews will be carried out as focus groups with three participants from each of the three counselling groups and a member of the research team.

Eligible participants will be assigned a group, with the first group starting in early 2025.

Measurements At baseline, before starting the first session of the program, the women will be asked to fill in questionnaires about their sociodemographic and background information and the following validated and standardized questionnaires; the Adult ADHD Self-Rating Scale (ASRS), the Generalized Anxiety Disorder assessment (GAD7), the Edinburg Postnatal Depression scale (EPDS), the Difficulties in Emotion Regulation Scale (DERS), and the Adult ADHD Quality of Life Measure (AAQoL). One week after the final 10-week program period, the women will be asked to fill in the following questionnaires: The Client Satisfaction Questionnaire (CSQ-8), the Credibility and Expectancy Scale (CEQ), the Negative Effects Questionnaire (NEQ) and again the six questionnaires that were also filled in at baseline. In addition to the quantitative measurements, we will conduct semi-structured interviews with three women from each group one week after the end of the program to assess their subjective perspectives on barriers and facilitators to participate in the program. We will use Clarke and Braun thematic analysis on the interview.

Statistical analysis plan Descriptive statistics For participant characteristics, we will summarize baseline sociodemographic and clinical characteristics using means and standard deviations for continuous variables, and frequencies and percentages for categorical variables. For program adherence, we will calculate adherence rates by assessing attendance records for each session.

Analyses For the primary outcomes, program satisfaction (CSQ-8), credibility and expectancy (CEQ), and negative effects (NEQ), we will summarize scores using means and standard deviations.

For the secondary outcomes, ADHD symptoms (ASRS), perceived stress (PSS), anxiety (GAD-7), depression (EPDS), emotion regulation (DERS-16), and quality of life (AAQoL), we will use paired t-test to compare pre- and post-intervention scores.

Power calculation Given the feasibility nature of this study, a formal power calculation is not conducted. However, the sample size of 30 participants, divided into three groups, is deemed sufficient to provide preliminary insights into program feasibility, adherence, and potential impacts on clinical outcomes.

Processing of personal data in the project All personal data will be processed in compliance with the General Data Protection Regulation (GDPR) and the Danish Data Protection Act. Any personally sensitive information is processed by OPEN (Open, Patient data Explorative Network) in personally identifiable form for as long as it is necessary for the research purpose. The storages of information are in accordance with responsible research practice and in relation to general data protection regulation. Individual participants will not be identifiable in published data, as the information of trial participants is anonymized, and individuals cannot be recognized. We will prioritize the protection of participants privacy and adhere to ethical guidelines. Anonymization involves removing personal identification details to prevent the disclosure of individual participants identities in published results and by reporting results that are based on at least 5 individuals. When the data is no longer necessary for the research project, it will be sent to the national archive and stored for five years. The project is registered at the University of Southern Denmark (journal nr: 12.303 - HELP - Mental health in pregnant women and new mothers with ADHD).

Economy The initiative for this trial was taken by associate professor Kathrine Bang Madsen. Funding is provided by Sygeforsikring "danmark" (Journalnr. 2021-0139 HELP - Mental health in pregnant women and new mothers with ADHD) as part of a larger project called HELP with an amount of DKK 5 mio, of which DKK 1.5 mio covers the development and evaluation of the counselling program. The financial support cover costs related to program development (to ADHD-foreningen), participant recruitment, and data analysis, and is administered by the University of Southern Denmark (SDU). The funding body has had no role in the study design, data collection, data analysis, data interpretation, or manuscript writing.

Recruitment and informed consent The Danish ADHD Association will advertise for the counselling program and the research project on their homepage and social media platforms. Those interested in participating can sign up by providing their email address via the homepage. They will then receive an email with details about the research project and are encouraged to reply with their phone number. The instructor of the program from the Danish ADHD Association will contact the participant by phone and screen the participant based on the eligibility criteria and provide the participant with information about the study. The verbal information given by phone includes the purpose and method of the program and the feasibility study, the voluntary nature of participation, that neither participation or non-participation will have an influence on other treatment options available to the individual, and the right to a consideration period (one week). The consent process is a dialogue, and the individual participant can ask questions about the program and study.

During the phone conversation, participants will be asked about their pregnancy status, since they will need to be pregnant. They are asked to share information about their ADHD diagnosis, including when they were diagnosed. Additionally, we will collect information about their living situation, such as whether they live with the child's father, their employment status, and similar details. If the participant meets the inclusion and exclusion criteria and decides to participate in the study, she will receive written information about the study and a consent form through e-mail via REDCap (Research Electronic Data Capture), which can be signed electronically. From the day of receiving the written information, the participant will have one week to consider participating. After signing, the participant will receive a copy of the consent form. The consent form will be stored in REDCap.

Ethics The trial poses minimal risks and offers potential therapeutic benefits that justify its conduct. The intervention is expected to significantly improve participants well-being and quality of life, benefiting both mother and baby. The counselling program AMOR is the first program to address the needs of pregnant women and new mothers. However, based on experiences with similar online programs for adults with ADHD (outside the perinatal period), the program is expected to enhance understanding of ADHD during pregnancy and childbirth, providing practical strategies for managing daily life during pregnancy and as a new parent. Other studies have not reported on negative effects, however, during each session, participants will be informed by the instructor to contact their general practitioner, midwife, or health nurse if they need more assistance than the program can provide. In addition, we will assess any potential negative effects after the end of the program. Participants will be informed of their rights and the compensation scheme for any injury related to the intervention.

Should participants exhibit scores exceeding 15 on the Generalized Anxiety Disorder-7 (GAD-7) scale and 18 on the Edinburgh Postnatal Depression Scale (EPDS) at baseline, they will be contacted by phone by one of the responsible investigators and encouraged to consult with their healthcare provider, such as their doctor or midwife and they will be informed that they are not eligible to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women or new mothers with an ADHD diagnosis (WHO ICD-10; F90 or F98.8)
* above 18 years
* access to a computer and the internet
* speaks and reads Danish

Exclusion Criteria:

* severe mental disorders, such as mental retardation, schizophrenia, psychosis or bipolar disorder
* a score above 15 on the Generalized Anxiety Disorder assessment or a score above 18 on the Edinburg Postnatal Depression scale administered
* current alcohol or substance abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2025-01-22 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
The Negative Effects Questionnaire (NEQ) | From enrollment to the end of the program 11 weeks
  Measure of experienced negative effects during treatment. It contains 20 items that are scored on a five-point Likert-scale (0-4) and differentiates between negative effects that are attributed to treatment and those possibly caused by other circumstances, as well as one open-ended questions.
The Credibility and Expectancy Scale (CEQ) | From enrollment to the end of the program 11 weeks
  Credibility of the intervention is measured by the third item from the Credibility and Expectancy Scale (CEQ): "How confident would you be in recommending this treatment to a friend who experiences similar problems?". Moreover, participants will be asked how likely they will be to continue to use the techniques from the program, with response options ranging from: "Very unlikely" to "Very likely".
Adherence | From enrollment to the end of the program
  Adherence is assessed by drop-out rates and participation in the sessions
The Client Satisfaction Questionare (CSQ-8) | From enrollment to the end of the program 11 weeks
  A measure of the participants' satisfaction with the intervention. The questionnaire consist of eight items measured on a four-point scale with total scores ranging from 8-32.

SECONDARY OUTCOMES:
The Adult ADHD Self-Rating Scale (ASRS) | From enrollment to the end of the program 11 weeks
  Designed to assess core symptoms of ADHD and includes 18 items rated on a five-point scale from: "Never" to "Very often".
The Perceived Stress Scale (PSS) | From enrollment to the end of the program 11 weeks
  Designed to assess the level of perceived stress during the past month. The scale includes 14 items and responses are rated on a five-point scale from "Never" to "Very often".
The Generalized Anxiety Disorder assessment (GAD7) | From enrollment to the end of the program 11 weeks
  Screens levels of anxiety and consists of 7 items scored on a 0-3 scale. While the GAD-7 was originally developed to measure generalized anxiety disorder, it has also been validated as a general measure of symptom severity of anxiety across different anxiety disorders in heterogeneous samples.
The Edinburg Postnatal Depression scale (EPDS) | From enrollment to the end of the program 11 weeks
  Questionnaire used worldwide to screen pregnant women and new mothers for depression in the perinatal period, translated, and validated in a Danish version. It is a ten-item questionnaire with sores ranging from 0-3.
The Difficulties in Emotion Regulation Scale - 16 item version (DERS-16) | From enrollment to the end of the program 11 weeks
  A self-report measure assessing individuals' typical levels of difficulties in emotion regulation.
The Adult ADHD Quality of Life Measure (AAQoL) | From enrollment to the end of the program 11 weeks
  Designed to assess quality of life during the past two weeks in adults with ADHD. AAQoL includes 29 items and responses are rated on a five-point scale from "Not at all/Never" to "Extremely/Very Often". The AAQoL yields a total score and four subscale scores: Life Productivity (eleven items), Psychological Health (six items), Life Outlook (seven items), Relationships (five items).

CONTACTS AND LOCATIONS:
Locations (1):
- The Danish ADHD Association, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young S, Emilsson B, Sigurdsson JF, Khondoker M, Philipp-Wiegmann F, Baldursson G, Olafsdottir H, Gudjonsson G. A randomized controlled trial reporting functional outcomes of cognitive-behavioural therapy in medication-treated adults with ADHD and comorbid psychopathology. Eur Arch Psychiatry Clin Neurosci. 2017 Apr;267(3):267-276. doi: 10.1007/s00406-016-0735-0. Epub 2016 Oct 17. PMID 27752827
- [Background] Nordby ES, Kenter RMF, Lundervold AJ, Nordgreen T. A self-guided Internet-delivered intervention for adults with ADHD: A feasibility study. Internet Interv. 2021 Jun 15;25:100416. doi: 10.1016/j.invent.2021.100416. eCollection 2021 Sep. PMID 34401375
- [Background] Brod M, Adler LA, Lipsius S, Tanaka Y, Heinloth AN, Upadhyaya H. Validation of the adult attention-deficit/hyperactivity disorder quality-of-life scale in European patients: comparison with patients from the USA. Atten Defic Hyperact Disord. 2015 Jun;7(2):141-50. doi: 10.1007/s12402-014-0160-z. Epub 2015 Jan 7. PMID 25563210
- [Background] Visted E, Solbakken OA, Maeland S, Fadnes LT, Bjerrum LB, Nordhus IH, Flo-Groeneboom E. Validation of a brief version of the Difficulties in Emotion Regulation Scale (DERS-16) with an older Norwegian population. Eur J Ageing. 2023 Jun 22;20(1):26. doi: 10.1007/s10433-023-00775-w. PMID 37347324
- [Background] Smith-Nielsen J, Matthey S, Lange T, Vaever MS. Validation of the Edinburgh Postnatal Depression Scale against both DSM-5 and ICD-10 diagnostic criteria for depression. BMC Psychiatry. 2018 Dec 20;18(1):393. doi: 10.1186/s12888-018-1965-7. PMID 30572867
- [Background] Lowe B, Decker O, Muller S, Brahler E, Schellberg D, Herzog W, Herzberg PY. Validation and standardization of the Generalized Anxiety Disorder Screener (GAD-7) in the general population. Med Care. 2008 Mar;46(3):266-74. doi: 10.1097/MLR.0b013e318160d093. PMID 18388841
- [Background] Beard C, Bjorgvinsson T. Beyond generalized anxiety disorder: psychometric properties of the GAD-7 in a heterogeneous psychiatric sample. J Anxiety Disord. 2014 Aug;28(6):547-52. doi: 10.1016/j.janxdis.2014.06.002. Epub 2014 Jun 14. PMID 24983795
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Kessler RC, Adler L, Ames M, Demler O, Faraone S, Hiripi E, Howes MJ, Jin R, Secnik K, Spencer T, Ustun TB, Walters EE. The World Health Organization Adult ADHD Self-Report Scale (ASRS): a short screening scale for use in the general population. Psychol Med. 2005 Feb;35(2):245-56. doi: 10.1017/s0033291704002892. PMID 15841682
- [Background] Rozental A, Kottorp A, Forsstrom D, Mansson K, Boettcher J, Andersson G, Furmark T, Carlbring P. The Negative Effects Questionnaire: psychometric properties of an instrument for assessing negative effects in psychological treatments. Behav Cogn Psychother. 2019 Sep;47(5):559-572. doi: 10.1017/S1352465819000018. Epub 2019 Mar 15. PMID 30871650
- [Background] Kajamaa A, Mattick K, de la Croix A. How to ... do mixed-methods research. Clin Teach. 2020 Jun;17(3):267-271. doi: 10.1111/tct.13145. Epub 2020 Feb 24. PMID 32092789
- [Background] Nimmo-Smith V, Merwood A, Hank D, Brandling J, Greenwood R, Skinner L, Law S, Patel V, Rai D. Non-pharmacological interventions for adult ADHD: a systematic review. Psychol Med. 2020 Mar;50(4):529-541. doi: 10.1017/S0033291720000069. Epub 2020 Feb 10. PMID 32036811
- [Background] Andersson A, Garcia-Argibay M, Viktorin A, Ghirardi L, Butwicka A, Skoglund C, Bang Madsen K, D'onofrio BM, Lichtenstein P, Tuvblad C, Larsson H. Depression and anxiety disorders during the postpartum period in women diagnosed with attention deficit hyperactivity disorder. J Affect Disord. 2023 Mar 15;325:817-823. doi: 10.1016/j.jad.2023.01.069. Epub 2023 Jan 18. PMID 36681302
- [Background] Attkisson CC, Zwick R. The client satisfaction questionnaire. Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval Program Plann. 1982;5(3):233-7. doi: 10.1016/0149-7189(82)90074-x. PMID 10259963
- [Background] Simon V, Czobor P, Balint S, Meszaros A, Bitter I. Prevalence and correlates of adult attention-deficit hyperactivity disorder: meta-analysis. Br J Psychiatry. 2009 Mar;194(3):204-11. doi: 10.1192/bjp.bp.107.048827. PMID 19252145
- [Background] Kittel-Schneider S, Quednow BB, Leutritz AL, McNeill RV, Reif A. Parental ADHD in pregnancy and the postpartum period - A systematic review. Neurosci Biobehav Rev. 2021 May;124:63-77. doi: 10.1016/j.neubiorev.2021.01.002. Epub 2021 Jan 28. PMID 33516734
- [Background] Anderson KN, Ailes EC, Danielson M, Lind JN, Farr SL, Broussard CS, Tinker SC. Attention-Deficit/Hyperactivity Disorder Medication Prescription Claims Among Privately Insured Women Aged 15-44 Years - United States, 2003-2015. MMWR Morb Mortal Wkly Rep. 2018 Jan 19;67(2):66-70. doi: 10.15585/mmwr.mm6702a3. PMID 29346342
- [Background] Song P, Zha M, Yang Q, Zhang Y, Li X, Rudan I; Global Health Epidemiology Reference Group (GHERG). The prevalence of adult attention-deficit hyperactivity disorder: A global systematic review and meta-analysis. J Glob Health. 2021 Feb 11;11:04009. doi: 10.7189/jogh.11.04009. PMID 33692893
- [Background] Young S, Adamo N, Asgeirsdottir BB, Branney P, Beckett M, Colley W, Cubbin S, Deeley Q, Farrag E, Gudjonsson G, Hill P, Hollingdale J, Kilic O, Lloyd T, Mason P, Paliokosta E, Perecherla S, Sedgwick J, Skirrow C, Tierney K, van Rensburg K, Woodhouse E. Females with ADHD: An expert consensus statement taking a lifespan approach providing guidance for the identification and treatment of attention-deficit/ hyperactivity disorder in girls and women. BMC Psychiatry. 2020 Aug 12;20(1):404. doi: 10.1186/s12888-020-02707-9. PMID 32787804
- [Background] Posner J, Polanczyk GV, Sonuga-Barke E. Attention-deficit hyperactivity disorder. Lancet. 2020 Feb 8;395(10222):450-462. doi: 10.1016/S0140-6736(19)33004-1. Epub 2020 Jan 23. PMID 31982036
- See also: Related Info — https://adhd.dk/kursus/help-raadgivningsforloeb-for-gravide/